CLINICAL TRIAL: NCT02246647
Title: Biomarkers for Intestinal Permeability in Patients With Functional Lower Gastrointestinal Disorders Associated With Constipation.
Brief Title: Biomarkers for Intestinal Permeability in Patients With Constipation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry)
Responsible Party: Principal Investigator, Madhusudan (Madhu) Grover, MBBS, Principal Investigator, Mayo Clinic
Other Study IDs: 14-002382
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2019-08-21 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Intestinal Diseases; Irritable Bowel Syndrome; Constipation
MeSH Terms: conditions — Intestinal Diseases; Irritable Bowel Syndrome; Constipation | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colonic Biopsies Duodenal Biopsies Blood Urine Fecal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy volunteers: Permeability measurement: Ingestion of saccharides {mannitol (regular, 12C) 100 mg, lactulose 1 g and labelled (13C mannitol) 100 mg} in 250ml of water Esophagogastroduodenoscopy Flexible sigmoidoscopy
  Interventions: Diagnostic Test: Permeability measurement; Procedure: Esophagogastroduodenoscopy; Procedure: Flexible sigmoidoscopy
- IBS-C: Permeability measurement: Ingestion of saccharides (mannitol (regular, 12C) 100 mg, lactulose 1 g and labelled (13C mannitol) 100 mg} in 250ml of water Esophagogastroduodenoscopy Flexible sigmoidoscopy
  Interventions: Diagnostic Test: Permeability measurement; Procedure: Esophagogastroduodenoscopy; Procedure: Flexible sigmoidoscopy

INTERVENTIONS:
Diagnostic Test: Permeability measurement — Saccharide excretion was compared between IBS-C and healthy volunteers
  Other Names: 12C Mannitol; 13C Mannitol; Lactulose
Procedure: Esophagogastroduodenoscopy — Duodenal biopsies were collected from IBS-C and healthy volunteers
Procedure: Flexible sigmoidoscopy — Colonic biopsies were collected from IBS-C and healthy volunteers

SUMMARY:
Our overall objective with this study is firstly to provide a comprehensive assessment of intestinal permeability, mucosal barrier function using existing biomarkers and secondly to explore novel biomarkers for measuring intestinal permeability in patients with constipation predominant Irritable Bowel Syndrome (IBS-C).

DETAILED DESCRIPTION:
In order to determine the differences in permeability in IBS-C in comparison with healthy volunteers, the following will be determined: differences in in vivo small intestinal and colonic permeability, differences in small intestinal and colonic mucosal barrier function, differences in effects of fecal supernatants on barrier function of T84 monolayers, and differences in novel biomarkers for intestinal permeability

ELIGIBILITY:
Inclusion criteria:

1. 18 - 65 years old
2. IBS-C by Rome III criteria (for IBS-C participants)
3. No abdominal surgery (except appendectomy and cholecystectomy)

Exclusion criteria:

1. History of Inflammatory Bowel Disease (IBD) , microscopic colitis or celiac disease
2. Use of tobacco products within the past 6 months
3. Use of NSAIDs or aspirin within the past week
4. Use of oral corticosteroids within the previous 6 weeks
5. Ingestion of artificial sweeteners such as Splenda (sucralose), Nutrasweet (aspartame), lactulose or mannitol 2 days before the study begins, e.g., foods to be avoided are sugarless gums or mints and diet soda
6. Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before study begins

   1. Any treatment specifically taken for IBS, including loperamide, cholestyramine, alosetron
   2. Drugs with a known pharmacological activity at 5-HT4, 5-HT2b or 5-HT3 receptors (e.g, tegaserod, ondansetron, tropisetron, granisetron, dolasetron, mirtazapine);
   3. All narcotics (e.g, codeine, morphine, and propoxyphene, either alone or in combination)
   4. Anti-cholinergic agents (e.g, dicyclomine, hyoscyamine, propantheline).
   5. Ultram
   6. GI preparations

      * Anti-nausea agents (e.g, trimethobenzamide, promethazine, prochlorperazine, dimenhydrinate, hydroxyzine)
      * Osmotic laxative agents (e.g, lactulose, sorbitol or PEG solutions as Miralax and Glycolax)
      * Prokinetic agents (e.g, cisapride, metoclopramide, itopride, domperidone);
   7. Antimuscarinics;
   8. Peppermint oil;
   9. Systemic antibiotics, rifaximin, metronidazole.
7. Bleeding disorders or medications that increase risk of bleeding from mucosal biopsies.
8. Score > 8 for anxiety or depression on Hospital anxiety and depression scale.
9. Pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBS-Constipation patients and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12-08 (Actual); Study Completion 2016-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhusudan Grover, MBBS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: Healthy subjects ages 18 - 65 Must not have had any abdominal surgeries, IBS, IBD, microscopic colitis or celiac disease. Must not have used tobacco products in the last 6 months. Must not have used corticosteroids in the last 6 weeks. Must not have taken any treatment specifically taken for IBS, including loperamide, cholestyramine, alosetron . Must not be taking any drugs with a known pharmacological activity at 5-HT4, 5-HT2b or 5-HT3 receptors. Must not have taken anti-cholinergic agents (e.g. dicyclomine, hyoscyamine, propantheline), Ultram. No GI preparations
  * Anti-nausea agents (e.g., trimethobenzamide, promethazine, prochlorperazine, dimenhydrinate, hydroxyzine)
  * Osmotic laxative agents (e.g, lactulose, sorbitol or PEG solutions as MiraLAX and GlycoLax) - Prokinetic agents (e.g, cisapride, metoclopramide, itopride, domperidone); Antimuscarinics;Peppermint oil;Systemic antibiotics, rifaximin, metronidazole. Must not have a bleeding disorder or medications that incr
- IBS-C: Age (yr) 18 to 65 Must have IBS-C by Rome III criteria No abdominal surgery (except appendectomy and cholecystectomy) Exclusion criteria: Must have no History of IBD (Crohn's disease or ulcerative colitis), microscopic colitis or celiac disease. Use of tobacco products within the past 6 months (since nicotine may affect intestinal permeability) Use of NSAIDs or aspirin within the past week (since NSAIDs affect intestinal permeability) Use of oral corticosteroids within the previous 6 weeks No Ingestion of artificial sweeteners such as SplendaTM (sucralose), NutraSweet TM(aspartame), lactulose or mannitol 2 days before the study begins, e.g., foods to be avoided are sugarless gums or mints and diet soda. Ingestion of any prescription, over the counter, or herbal medications which can affect gastrointestinal transit 7 days before study begins ny treatment specifically taken for IBS, including loperamide, cholestyramine, alosetron No drugs with a known pharmacological activity at 5
Period: Overall Study
Arm/Group | Healthy Volunteers | IBS-C
Started | 19 | 20
Completed (2 subjects (1 in Healthy Volunteers and 1 in IBS-C) would count as screen failures & hence withdrawn) | 18 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Healthy Volunteers: Healthy volunteers between ages 18 - 65, who have not history of IBS.
- IBS-C: Volunteers who have been diagnosed with IBS - Constipation (IBS-C)
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | IBS-C | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.37 (2.82) | 43.06 (2.78) | 44.24 (1.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18 | 19 | 37

OUTCOME MEASURES:

1. Primary Outcome: Lactulose:C13 Mannitol Excretion Ratio 8-24hrs.
Description: In vivo measurement of intestinal permeability using 13C mannitol & lactulose was used. High performance liquid chromatography-tandem mass spectrometry was used to measure concentrations calculated using the overall urine volume excreted in each interval. Concentrations of 13C adjusted for the % of 13C in 12C mannitol (4.98% of 12C mannitol excreted was subtracted from 13C mannitol values; determined by analyzing replicate samples of control urine). All lactulose or 13C mannitol concentrations 8-24hr post-ingestion were used to determine colonic permeability. Lactulose to 13C mannitol excretion ratios, as a measure of dose of saccharide administered, were calculated.
Time Frame: 8-24 hr post test-dose administration
Measure: Mean (Standard Error); unit: Ratio
Groups:
- Healthy Volunteers: Ingestion of saccharides (mannitol (regular, 12C) 100 mg, lactulose 1 g and (non-radioactive) 13C labeled mannitol, 100 mg and sucralose, 50 mg) in 250ml of water Esophagogastroduodenoscopy Flexible sigmoidoscopy
  Esophagogastroduodenoscopy: Duodenal biopsies will be collected from Healthy Volunteers.
  Flexible sigmoidoscopy: Colonic biopsies will be collected from Healthy Volunteers.
- IBS - C: Ingestion of saccharides (mannitol (regular, 12C) 100 mg, lactulose 1 g and (non-radioactive) 13C labeled mannitol, 100 mg and sucralose, 50 mg) in 250ml of water Esophagogastroduodenoscopy Flexible sigmoidoscopy
  Esophagogastroduodenoscopy: Duodenal biopsies will be collected from IBS - C cases.
  Flexible sigmoidoscopy: Colonic biopsies will be collected from IBS - C cases.
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 18 | 19
Ratio | 0.01 (0.004) | 0.02 (0.005)
Statistical Analysis 1: Comparison: Healthy Volunteers vs IBS - C; Test type: Other; p = 0.87, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.01

2. Secondary Outcome: Lactose:C13 Mannitol Excretion Ratio 0-2hours
Time Frame: 0-2 hr post-test dose administration
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 18 | 19
Ratio | 0.007 (0.0004) | 0.01 (0.001)

3. Secondary Outcome: Baseline Transmucosal Resistance (TMR) of Duodenal Mucosa
Time Frame: Baseline
Population: Two participants ( 1 in Healthy volunteers and 1 in IBS-C ) were not analysed for the Baseline transmucosal resistance (TMR) of duodenal mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure etc.
Measure: Mean (Standard Error); unit: Ω*sq.cm
Groups:
- Healthy Volunteers: Four biopsies from duodenum from the Healthy Volunteers were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran.
- IBS - C: Four biopsies from duodenum from the IBS - C cases were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 17 | 18
Ω*sq.cm | 29.8 (1.94) | 28.16 (1.96)

4. Secondary Outcome: Cumulative FITC-Dextran (4kDa) Concentration Across Duodenal Mucosa
Description: This is not a pharmacokinetic or pharmacodynamic measure. Hence only one time assessment is made 3 hours after FITC-Dextran (4kDa) administration.
Time Frame: 3 hours post FITC-Dextran (4kDa) administration
Population: Four participants (2 in Healthy volunteers and 2 in IBS-C) were not analysed for the Cumulative FITC-Dextran (4kDa) concentration across duodenal mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: ng/mL
Groups:
- Healthy Volunteers: Four biopsies from each site from the Healthy Volunteers were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran.
- IBS - C: Four biopsies from each site from the IBS - C cases were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 17
ng/mL | 123.3 (24.29) | 156.8 (33.73)

5. Secondary Outcome: Rate of FITC-Dextran (4kDa) Flux Across Duodenal Mucosa
Description: as for outcome 4
Time Frame: Over 3 hours post FITC-Dextran (4kDa) administration
Population: Four participants ( 2 in Healthy volunteers and 2 in IBS-C ) were not analysed for the Rate of FITC-Dextran (4kDa) flux across duodenal mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure etc.
Measure: Mean (Standard Error); unit: ng/hr/sq.cm
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 17
ng/hr/sq.cm | 4980 (1044) | 6528 (1584)

6. Secondary Outcome: Baseline Transmucosal Resistance (TMR) of Colonic Mucosa
Time Frame: Baseline
Population: One participant in IBS-C was not analysed for the Baseline Transmucosal Resistance (TMR) of Colonic Mucosa due to various reasons such inadequate size of the biopsy specimen.
Measure: Mean (Standard Error); unit: Ω*sq.cm
Groups:
- Healthy Volunteers: Four biopsies from colon from the Healthy Volunteers were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran.
- IBS - C: Four biopsies from colon from the IBS - C cases were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured.Average TMR and Isc across 3-4 biopsies/subject were calculated.Paracellular flux across biopsies was measured using 4 kDa FITC-Dextran administered on the mucosal side (1 mg/mL chamber concentration). Cumulative flux at the end of three hours and rate of flux was calculated for FITC-Dextran
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 18 | 18
Ω*sq.cm | 17.60 (1.70) | 19.06 (1.10)

7. Secondary Outcome: Cumulative FITC-Dextran (4kDa) Concentration Across Colonic Mucosa
Time Frame: 3 hours post FITC-Dextran (4kDa) administration
Population: 7 participants (2 in Healthy volunteers and 5 in IBS-C) were not analysed for the Cumulative FITC-Dextran (4kDa) Concentration Across Colonic Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 14
ng/mL | 132.2 (24.23) | 122.5 (27.44)

8. Secondary Outcome: Rate of FITC-Dextran (4kDa) Flux Across Colonic Mucosa
Time Frame: Over 3 hours post FITC-Dextran (4kDa) administration
Population: 7 participants (2 in Healthy volunteers and 5 in IBS-C) were not analysed for the Rate of FITC-Dextran (4kDa) Flux Across Colonic Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: ng/hr/sq.cm
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 14
ng/hr/sq.cm | 4931 (1156) | 6069 (1030)

9. Secondary Outcome: Cumulative E.Coli Bio- Particle K12 Concentration Across Duodenal Mucosa
Time Frame: 3 hours post E.coli Bio- Particle administration
Population: 11 participants (4 in Healthy volunteers and 7 in IBS-C) were not analysed for Cumulative E.Coli Bio- Particle K12 Concentration Across Duodenal Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: CFU/ml
Groups:
- Healthy Volunteers: Four biopsies from duodenum from the Healthy Volunteers were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured. Average TMR and Isc across 3-4 biopsies/subject were calculated. Transcellular transport was studied by using translocation of the fluorescently labeled E. coli K-12 Bio-Particles was measured using a 107 CFU/mL chamber concentration on the mucosal side. Cumulative flux at the end of three hours and rate of flux was calculated for E. coli K-12 Bio-Particles.
- IBS - C: Four biopsies from duodenum from the IBS - C cases were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured. Average TMR and Isc across 3-4 biopsies/subject were calculated. Transcellular transport was studied by using translocation of the fluorescently labeled E. coli K-12 Bio-Particles was measured using a 107 CFU/mL chamber concentration on the mucosal side. Cumulative flux at the end of three hours and rate of flux was calculated for E. coli K-12 Bio-Particles.
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 14 | 12
CFU/ml | 1.48*10^4 (2.6*10^3) | 1.82*10^4 (6.0*10^3)

10. Secondary Outcome: Rate of E.Coli Bio- Particle K12 Flux Across Duodenal Mucosa
Time Frame: Over 3 hours post E.coli Bio- Particle administration
Population: 11 participants (4 in Healthy volunteers and 7 in IBS-C) were not analysed for Rate of E.Coli Bio- Particle K12 Flux Across Duodenal Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: CFU/h/sq.cm
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 14 | 12
CFU/h/sq.cm | 5.42*10^5 (1.2*10^5) | 5.70*10^5 (1.90*10^5)

11. Secondary Outcome: Cumulative E.Coli Bio- Particle K12 Concentration Across Colonic Mucosa
Time Frame: 3 hours post E.coli Bio- Particle administration
Population: 7 participants (2 in Healthy volunteers and 5 in IBS-C) were not analysed for Cumulative E.coli Bio- Particle K12 Concentration Across Colonic Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: CFU/ml
Groups:
- Healthy Volunteers: Four biopsies from colon from the Healthy Volunteers were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured. Average TMR and Isc across 3-4 biopsies/subject were calculated. Transcellular transport was studied by using translocation of the fluorescently labeled E. coli K-12 Bio-Particles was measured using a 107 CFU/mL chamber concentration on the mucosal side. Cumulative flux at the end of three hours and rate of flux was calculated for E. coli K-12 Bio-Particles.
- IBS - C: Four biopsies from colon from the IBS - C cases were mounted in 4 mL Ussing chambers (Physiologic Instruments, San Diego, CA, USA) exposing 0.031 sq.cm area, within 45 min of collection. Chambers were filled with Krebs with 10 mM mannitol (mucosal side) and Krebs with 10 mM glucose (submucosal side).Baseline transmucosal resistance (TMR) and short circuit current (Isc) of each tissue was measured. Average TMR and Isc across 3-4 biopsies/subject were calculated. Transcellular transport was studied by using translocation of the fluorescently labeled E. coli K-12 Bio-Particles was measured using a 107 CFU/mL chamber concentration on the mucosal side. Cumulative flux at the end of three hours and rate of flux was calculated for E. coli K-12 Bio-Particles.
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 14
CFU/ml | 1.07*10^4 (1.8*10^3) | 2.09*10^4 (6.8*10^3)

12. Secondary Outcome: Rate of E.Coli Bio- Particle K12 Flux Across Colonic Mucosa
Time Frame: Over 3 hours post E.coli Bio- Particle administration
Population: 7 participants (2 in Healthy volunteers and 5 in IBS-C) were not analysed for Rate of E.Coli Bio- Particle K12 Flux Across Colonic Mucosa due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: CFU/h/sq.cm
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 14
CFU/h/sq.cm | 4.26*10^5 (5.3*10^4) | 7.67*10^5 (4.19*10^5)

13. Secondary Outcome: Duodenal Impedance
Time Frame: Baseline
Population: 12 participants (2 in Healthy volunteers and 10 in IBS-C) were not analysed for Duodenal impedance due to various reasons such inadequate size of the biopsy specimen, participant did not show up for the procedure, etc.
Measure: Mean (Standard Error); unit: Ω
Groups:
- Healthy Volunteers: Volunteers fasted for eight hours and underwent sedated esophagogastroduodenoscopy. Duodenal impedance measurements were performed using a endoscopically passed catheter that measures electrical impedance of the duodenal epithelium by mucosal contact under direct visualization. A 2 mm diameter catheter was used with two 360° circumferential sensors placed at a separation of 2mm with the end of the distal ring being 1mm away from the catheter tip. The electrodes were connected to an impedance voltage transducer via thin wires, which ran the length of the catheter traversing through the working channel of the upper endoscope. The voltage generated by the transducer was limited to produce 10µA current at a frequency of 2 kHz. Impedance was measured every 90° in duodenal circumference with a decompressed lumen after suctioning of all fluid from the lumen. The catheter was embedded in the mucosa parallel to the two sensors and measurements were taken from a steady baseline for >10s.
- IBS - C: IBS - C cases fasted for eight hours and underwent sedated esophagogastroduodenoscopy. Duodenal impedance measurements were performed using a endoscopically passed catheter that measures electrical impedance of the duodenal epithelium by mucosal contact under direct visualization. A 2 mm diameter catheter was used with two 360° circumferential sensors placed at a separation of 2mm with the end of the distal ring being 1mm away from the catheter tip. The electrodes were connected to an impedance voltage transducer via thin wires, which ran the length of the catheter traversing through the working channel of the upper endoscope. The voltage generated by the transducer was limited to produce 10µA current at a frequency of 2 kHz. Impedance was measured every 90° in duodenal circumference with a decompressed lumen after suctioning of all fluid from the lumen. The catheter was embedded in the mucosa parallel to the two sensors and measurements were taken from a steady baseline for >10s.
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 16 | 9
Ω | 705.9 (42.73) | 729.5 (64.85)

14. Secondary Outcome: Mean Serum Endotoxin (Bacterial LPS) Levels
Time Frame: Fasting, one time measurement after 8 hours
Population: 2 participants (1 in healthy volunteers and 1 in IBS-C) were not analysed for Mean Serum Endotoxin (Bacterial LPS) Levels due to various reasons such as non-availability of the blood sample, technical errors, etc.
Measure: Mean (Standard Error); unit: EU/mL
Groups:
- Healthy Volunteers: Fasting, EDTA anti-coagulated, whole blood was collected from Healthy Volunteers. Samples were analyzed using an EAA kit (Spectral Diagnostic Inc, Toronto, Ontario, Canada) that utilizes a monoclonal IgM antibody specific for gram-negative bacterial lipopolysaccharide (LPS). Samples were tested in duplicate within one hour of collection using a Berthold SmartLine luminometer (photon-counting). The endotoxin activity level was calculated as follows: chemiluminescence (test sample-negative control)/chemiluminescence (positive-negative control). Average values for each participant were expressed as absolute units.
- IBS - C: Fasting, EDTA anti-coagulated, whole blood was collected from IBS - C cases. Samples were analyzed using an EAA kit (Spectral Diagnostic Inc, Toronto, Ontario, Canada) that utilizes a monoclonal IgM antibody specific for gram-negative bacterial lipopolysaccharide (LPS). Samples were tested in duplicate within one hour of collection using a Berthold SmartLine luminometer (photon-counting). The endotoxin activity level was calculated as follows: chemiluminescence (test sample-negative control)/chemiluminescence (positive-negative control). Average values for each participant were expressed as absolute units.
Arm/Group | Healthy Volunteers | IBS - C
Number analyzed (Participants) | 17 | 18
EU/mL | 0.35 (0.02) | 0.36 (0.03)

ADVERSE EVENTS:
Time Frame: 15 months-from the first participant screening to the last participants completion date
Groups:
- Healthy Volunteer: Healthy volunteers between ages 18 - 65, who have no history of IBS.
- IBS-C: ROME III IBS-C patients
Arm/Group | Healthy Volunteer | IBS-C
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Volunteer (N=18) | IBS-C (N=19)
Indigestion/Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) — Indigestion/Heartburn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less